CLINICAL TRIAL: NCT05755581
Title: Efficacy of Endocrine Therapy Compared to Chemotherapy as a Neoadjuvant Treatment for Patients With Hormone Receptor-positive and HER2-negative Breast Cancer.
Brief Title: Efficacy of Neoadjuvant Endocrine Therapy Compared to Chemotherapy in Breast Cancer Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Amal Ali Omar, Assistant lecturer, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Soh-Med-23-02-16
Record Dates: First submitted 2023-02-15; First posted 2023-03-06 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-02

CONDITIONS: Female Breast Cancer
Keywords: Neoadjuvant endocrine therapy ,neoadjuvant chemotherapy
MeSH Terms: interventions — Antineoplastic Agents, Hormonal

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into two groups:
  The first group (Arm A) will receive NCT; (Any approved Chemotherapy protocol by guidelines.
  The second group(Arm B) will receive NET; GnRH analog Goserelin acetate 3.6 mg every 4 weeks with tamoxifen 20 mg daily for premenopausal patients or an aromatase inhibitor for postmenopausal patients.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neoadjuvant chemotherapy group (Active Comparator): Patients in this arm will receive neoadjuvant chemotherapy as usual
  Interventions: Drug: Chemotherapy drug
- Neoadjuvant endocrine therapy group (Active Comparator): Patients in this group will receive neoadjuvant endocrine therapy
  Interventions: Drug: Hormonal Antineoplastics

INTERVENTIONS:
Drug: Hormonal Antineoplastics — the Neoadjuvant endocrine therapy group will receive neoadjuvant hormonal therapy.
  Arms: Neoadjuvant endocrine therapy group
Drug: Chemotherapy drug — the Neoadjuvant chemotherapy group will receive neoadjuvant chemotherapy.
  Arms: Neoadjuvant chemotherapy group

SUMMARY:
Eligible patients will be divided into two groups; one will receive neoadjuvant endocrine therapy and the other one will receive neoadjuvant chemotherapy.

DETAILED DESCRIPTION:
Patients will be randomized into two groups:

The first group (Arm A) will receive NCT; (Any approved Chemotherapy protocol by guidelines.

The second group(Arm B) will receive NET; GnRH analog Goserelin acetate 3.6 mg every 4 weeks with tamoxifen 20 mg daily for premenopausal patients or an aromatase inhibitor for postmenopausal patients.

* Before and during treatments (every 3 weeks for the NCT group, and every 4 weeks for the NET group), the clinical assessment will be performed for all patients.
* All patients will undergo breast magnetic resonance imaging (MRI) before the start of treatment, after 12 weeks (3 months) of treatment, and after the end of treatment before surgery.
* We will determine the objective tumor response with every measurement method and assess the response according to the Response Evaluation Criteria in Solid Tumor (RECIST) version 1.1.
* Treatment will be continued for 19-21 weeks before surgery for the chemotherapy group and 24 weeks for the endocrine therapy group.
* Ki-67 will be assessed using a sample of the core biopsy before treatment and a surgery specimen after treatment.
* Adverse events will be recorded at every patient visit and will be assessed according to the Common Terminology Criteria for Adverse Events Version 5.0.
* Surgery will be performed between the 24th and 26th week.
* Arm B Patients who will develop PD or SD after 6 months of treatment will be shifted to arm A.

The primary endpoint will be;

* The clinical response rate at the end of neoadjuvant treatment, as will be determined using caliper and MRI measurements.
* A clinical response included either a complete response (CR), a partial response (PR), Progressive Disease (PD), or Stable Disease (SD) according to the (RECIST) version 1.1.

Secondary endpoints will be;

* The rate of pathological complete response (pCR).
* The rate of breast conservation surgery.
* Ki-67 changes.
* The length of time to maximum response within a treatment period.
* The Adverse events associated with each treatment arm.

ELIGIBILITY:
Inclusion Criteria:

* Any histological type of invasive breast cancer. All grades of breast cancer (I, II, III). ER-positive and/or PR-positive, HER2-negative breast cancer. ER and/or PR level of positivity ≥34 % (score 4 according to modified Allred score).

Clinical Stages: any T N1-3, or T2-4 any N, M0.

Exclusion Criteria:

* Hormone receptor positivity < 34%. inflammatory breast cancer Metastatic breast cancer. Recurrent breast cancer. Other malignancy. Unfit patients for chemotherapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Clinical response rate | 6 months
  The primary endpoint will be; The clinical response rate at the end of neoadjuvant treatment, as will be determined using caliper and MRI measurements according to the (RECIST) version 1.1.

SECONDARY OUTCOMES:
pathological complete response | 6 months
  The rate of pathological complete response after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Amal Ali, MD, Principal Investigator — Assistant lecturer
Locations (1):
- amal Ali, Sohag, Egypt